CLINICAL TRIAL: NCT03421639
Title: A Controlled Trial on Adenomyosis Treatment Comparing Aromatase Inhibitor Plus GnRH Analogue Versus GnRH Analog Alone
Brief Title: Aromatase Plus GnRH Analogue Versus GnRH Analog Alone in Adenomyosis
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre for Endocrinology and Reproductive Medicine, Italy (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR-01-18
Record Dates: First submitted 2018-01-30; First posted 2018-02-05 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Uterine Adenomyosis; Recurrent Implantation Failure; Menstrual Pain
Keywords: Implantation failure; Adenomyosis; increased uterine size; IVF; egg donation cycle
MeSH Terms: conditions — Adenomyosis; Dysmenorrhea | interventions — Gonadotropin-Releasing Hormone; Leuprolide; Control Groups; Aromatase Inhibitors; Aromatase

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial in two arms study (150 each one)
Who Masked: Participant, Care Provider
Masking Description: Patients will take similar kind medications by an indipendent person
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GnRH analog alone (Active Comparator): control group treated with GnRH analog alone
  Interventions: Drug: GnRH analog (11.25mg Leuprolide acetate)
- Aromatase inhibitor plus GnRH analog (Experimental): experimental group treated with aromatase inhibitor plus GnRH analog
  Interventions: Drug: Aromatase inhibitor and GnRH analog; Drug: Aromatase and GnRH analog (11.25mg Leuprolide acetate)

INTERVENTIONS:
Drug: GnRH analog (11.25mg Leuprolide acetate) — 11.25 Leuprolide acetate only one administration
  Other Names: Control group
  Arms: GnRH analog alone
Drug: Aromatase inhibitor and GnRH analog — 1mg/day of Anastrazole for 3 months
  Other Names: experimental group
  Arms: Aromatase inhibitor plus GnRH analog
Drug: Aromatase and GnRH analog (11.25mg Leuprolide acetate) — Leuprolide acetate 11.25mg only one
  Other Names: experimental group
  Arms: Aromatase inhibitor plus GnRH analog

SUMMARY:
With this study the investigators want to test which is the best medical treatment for symptomatic adenomyosis affecting women undergoing IVF and with previous implantation failure, between Aromatase inhibitor plus GnRH analog versus GnRH alone, in term pregnancy rate and uterine volume reduction.

DETAILED DESCRIPTION:
Recently it has been shown that adenomyosis negatively affects the pregnancy rate in IVF cycles. The investigators used in the past for the treatment of other benign gynecological diseases such as endometriosis and uterine myomas a combined therapy with Aromatase inhibitor plus GnRH analog. With this study the investigators want evaluate which is the best way to treat adenomyosis in order to obtain a higher pregnancy rate in women with symptomatic adenomyosis undergoing IVF who failed a previous IVF attempt. For these reasons the investigators set this controlled trial between GnRH analog plus Aromatase Inhibitor (3.75 mg monthly of Leuprolide plus 1.0mg day of Anastrazole for 3 months) versus an active comparator as GnRH analog alone (3.75 mg monthly of Leuprolide for 3 months) after the treatment patients will undergo embryo transfer of a cryopreserved blastocyst in a previous IVF cycle, and will be followed up for uterine dimension reduction and pain symptom reduction.

ELIGIBILITY:
Inclusion Criteria:

* women with healty conditions
* Adenomyosis
* increased uterine dimensions
* recurrent implantation failure

Exclusion Criteria:

* presence of systemic diseases

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
pregnancy after embryo transfer | 12 months
  after treatment patients undergo embryo transfer of a cryopreservad blastocyst

SECONDARY OUTCOMES:
uterine volume reduction | 12 months
  differences in uterine volume pre and post treatment evaluated by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: MARCO SBRACIA, MD, Study Chair — CERM-HUNGARIA
Locations (3):
- Spitali Amerikan, Tirana, Albania
- Nadezda Women's Health Hospital, Sofia, Bulgaria
- Cerm-Hungaria, Rome, Italy

IPD SHARING:
Plan to Share IPD: No